CLINICAL TRIAL: NCT00536874
Title: A Phase II Study of Neoadjuvant Gemcitabine and Oxaliplatin in Patients With Potentially Resectable Previously Untreated Pancreatic Adenocarcinoma
Brief Title: Gemcitabine and Oxaliplatin in Treating Patients With Pancreatic Cancer That Can Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-113; MSKCC-07113
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Results first posted 2015-12-17 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage IA pancreatic cancer; stage IB pancreatic cancer; stage IIA pancreatic cancer; stage IIB pancreatic cancer; stage III pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Oxaliplatin; Chemotherapy, Adjuvant; Neoadjuvant Therapy

ARMS (1):
- Gemcitabine And Oxaliplatin (Experimental): A Phase II Study of Neoadjuvant Gemcitabine And Oxaliplatin In Patients With Potentially Resectable Previously Untreated Pancreatic Adenocarcinoma
  Interventions: Drug: gemcitabine hydrochloride; Drug: oxaliplatin; Genetic: protein expression analysis; Genetic: proteomic profiling; Other: diagnostic laboratory biomarker analysis; Procedure: adjuvant therapy; Procedure: neoadjuvant therapy; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: gemcitabine hydrochloride — 1,000 mg/m2 IV over 100 minutes on day 1 every 14 days for 4 cycles
Drug: oxaliplatin — 80 mg/m2 IV over 2 hours on day 1 every 14 days for 4 cycles.
Genetic: protein expression analysis
Genetic: proteomic profiling
Other: diagnostic laboratory biomarker analysis
Procedure: adjuvant therapy
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving chemotherapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with oxaliplatin works in treating patients with pancreatic cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the overall 18-month survival of patients with radiographically resectable pancreatic adenocarcinoma treated with neoadjuvant gemcitabine and oxaliplatin followed by surgical resection and adjuvant gemcitabine.

Secondary

* To determine the safety, toxicity, and feasibility of this regimen in the neoadjuvant setting.
* To determine the feasibility of obtaining preoperative core tissue biopsies and the ability to use these biopsies to establish pathologic correlates of response following neoadjuvant therapy and to determine if xenografts can be developed from these core tissues.
* To determine the specific tumor marker response (CEA and CA19-9) to neoadjuvant therapy.
* To determine the prognostic accuracy of serum protein profiles in these patients.
* To determine the overall survival and patterns of tumor recurrence (local vs distant).

OUTLINE:

* Neoadjuvant therapy: Patients receive gemcitabine IV over 100 minutes and oxaliplatin IV over 2 hours on day 1. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity.
* Surgery: Within 2-6 weeks after completion of neoadjuvant therapy, patients undergo a laparoscopy that includes a pancreaticoduodenectomy or distal pancreatectomy with or without splenectomy.
* Adjuvant therapy: Beginning 4-16 weeks after surgery, patients receive gemcitabine IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 5 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo tumor tissue and blood sample collection periodically for correlative studies. Samples are analyzed for protein expression and tumor markers (CEA and CA19-9) pre- and post-neoadjuvant therapy via proteomic analysis. Tumor tissue samples are also banked for research purposes.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed pancreatic adenocarcinoma

  * No histology other than adenocarcinoma (e.g., neuroendocrine cancer or acinar cancer)

    * Patients with adenosquamous variants are eligible
* Radiographically resectable pancreatic cancer, as determined by a surgical oncologist

  * No metastatic or locally unresectable pancreatic adenocarcinoma
* No evidence of distant metastases by CT scan

  * Negative or pending laparoscopy for distant metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 4.0 mg/dL (if > 3.0, stented and known to be declining)
* Serum creatinine ≤ 1.6 mg/dL
* INR < 1.5 (therapeutic INR is allowed for patients receiving therapeutic anticoagulation)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study therapy
* No active infection, except for resolving cholangitis, that would preclude study enrollment

  * Neoadjuvant therapy may only be initiated when acute cholangitis has resolved
* No other malignancy within the past 3 years except for curatively treated basal cell carcinoma of the skin, cervical intraepithelial neoplasia, or localized prostate cancer with a PSA of < 5.0 ng/mL within ≥ 4 weeks of study entry (other circumstances with a recent concurrent or active malignancy will be adjudicated on a case-by-case basis by the principle investigator [PI] or co-PI)
* No known hypersensitivity to any of the components of oxaliplatin or gemcitabine
* No hypersensitivity to CT scan IV contrast dye not suitable for premedication
* No peripheral neuropathy ≥ grade 2
* No known HIV or hepatitis B or C infection (active, previously treated, or both)
* No other medical condition, including mental illness or substance abuse that, deemed by the investigator, would preclude study participation

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to > 25% of bone marrow
* More than 30 days since prior and no other concurrent investigational therapy
* No other prior therapy for pancreatic cancer
* No other concurrent chemotherapy, immunotherapy, or radiotherapy during neoadjuvant therapy
* Concurrent low molecular weight heparin or warfarin, where medically indicated, allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-10; Primary Completion 2012-09 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eileen O'Reilly, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Peter J. Allen, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] O'Reilly EM, Perelshteyn A, Jarnagin WR, Schattner M, Gerdes H, Capanu M, Tang LH, LaValle J, Winston C, DeMatteo RP, D'Angelica M, Kurtz RC, Abou-Alfa GK, Klimstra DS, Lowery MA, Brennan MF, Coit DG, Reidy DL, Kingham TP, Allen PJ. A single-arm, nonrandomized phase II trial of neoadjuvant gemcitabine and oxaliplatin in patients with resectable pancreas adenocarcinoma. Ann Surg. 2014 Jul;260(1):142-8. doi: 10.1097/SLA.0000000000000251. PMID 24901360

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine And Oxaliplatin: A Phase II Study of Neoadjuvant Gemcitabine And Oxaliplatin In Patients With Potentially Resectable Previously Untreated Pancreatic Adenocarcinoma
  gemcitabine hydrochloride: 1,000 mg/m2 IV over 100 minutes on day 1 every 14 days for 4 cycles
  oxaliplatin: 80 mg/m2 IV over 2 hours on day 1 every 14 days for 4 cycles.
  protein expression analysis
  proteomic profiling
  diagnostic laboratory biomarker analysis
  adjuvant therapy
  neoadjuvant therapy
  therapeutic conventional surgery
Period: Overall Study
Arm/Group | Gemcitabine And Oxaliplatin
Started | 39
Completed | 35
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine And Oxaliplatin
Number analyzed (Participants) | 39
Age, Continuous [Median (Standard Deviation); unit: years] | 63.5 (33.23401872)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at 18 Months
Description: Percentage of participants that were alive or survived at 18 months after randomization
Time Frame: 18 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemcitabine And Oxaliplatin
Number analyzed (Participants) | 35
percentage of participants | 63 [45 to 76]

2. Secondary Outcome: Overall Survival (Follow-Up Time)
Time Frame: From Baseline until 2 Years and Follow-Up, up to 120 months
Measure: Median (Full Range); unit: months
Arm/Group | Gemcitabine And Oxaliplatin
Number analyzed (Participants) | 35
months | 39.6 [12.3 to 57.7]

3. Secondary Outcome: Specific Tumor Marker Response (CEA) to Neoadjuvant Therapy
Time Frame: Baseline and 2 years
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Gemcitabine And Oxaliplatin
Number analyzed (Participants) | 35
ng/ml
  CEA (Pre-Therapy) | 4.2 [0.8 to 149]
  CEA (Post-Therapy) | 4.2 [0.8 to 82]

4. Secondary Outcome: RECIST Radiologic Response to Neoadjuvant Therapy
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR)=CR +PR
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Gemcitabine And Oxaliplatin
Number analyzed (Participants) | 35
participants
  Partial Response | 4
  Stable Disease | 28
  Progression of Disease | 3
  Inevaluable | 3

5. Secondary Outcome: Specific Tumor Marker Response (Ca 19-9) to Neoadjuvant Therapy
Time Frame: Baseline and 2 years
Measure: Median (Full Range); unit: U/ml
Arm/Group | Gemcitabine And Oxaliplatin
Number analyzed (Participants) | 35
U/ml
  Ca 19-9 (Pre-Therapy) | 133 [3 to 3816]
  Ca 19-9 (Post-Therapy) | 132 [5 to 2483]

6. Secondary Outcome: Specific Tumor Marker Response (CEA) to Neoadjuvant Therapy
Description: Percentage change in specific tumor marker (Carcinoembryonic antigen, CEA) levels in response to neoadjuvant therapy
Time Frame: Baseline and 2 years
Measure: Median (Full Range); unit: percent change
Arm/Group | Gemcitabine And Oxaliplatin
Number analyzed (Participants) | 35
percent change | -5.1 [-68 to 203]

7. Secondary Outcome: Specific Tumor Marker Response (Ca 19-9) to Neoadjuvant Therapy
Description: Percent change in specific tumor marker (Cancer Antigen 19-9, Ca 19-9) levels in response to neoadjuvant therapy
Time Frame: Baseline and 2 years
Measure: Median (Full Range); unit: percent change
Arm/Group | Gemcitabine And Oxaliplatin
Number analyzed (Participants) | 35
percent change | -25.6 [-85 to 289]

ADVERSE EVENTS:
Arm/Group | Gemcitabine And Oxaliplatin
Serious Adverse Events (participants affected / at risk) | 25/39
Other Adverse Events (participants affected / at risk) | 25/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine And Oxaliplatin (N=39)
Allergic reaction-Hypersensitivity (Immune system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Ascites (non-malignant) (Gastrointestinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
General disorder (General disorders) | 1 (1)
Sudden death (General disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 6 (6)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Anemia (Hemoglobin decrease) (Blood and lymphatic system disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Biliary tract infection (Infections and infestations) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bladder infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Infections and infestations -other (Infections and infestations) | 2 (2)
Injection site reaction (General disorders) | 1 (1)
Pancreatic anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine And Oxaliplatin (N=39)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Alkaline phosphatase increased (Investigations) | 2 (2)
Fatigue (General disorders) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 9 (9)
White blood cell decreased (Investigations) | 8 (8)
Lymphocyte count decreased (Investigations) | 5 (5)
Nausea (Gastrointestinal disorders) | 3 (3)
Neutrophil count decreased (Investigations) | 9 (9)
Abdominal pain (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes